CLINICAL TRIAL: NCT06531421
Title: Use of Equity Report Cards to Mitigate Disparities in Emergency Medical Services (EMS) Care for Injured Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: American Academy of Pediatrics (Other); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 00001103
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Pain, Acute
Keywords: Racial Groups
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: This is a pragmatic single-arm trial using an interrupted time-series design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Distribution of Equity Report Cards
  Interventions: Other: Equity Report Cards

INTERVENTIONS:
Other: Equity Report Cards — At month 2 the investigators will distribute EMS Agency-level 'Equity Report Cards' to both agency leadership and all frontline EMS providers. This 'Equity Report Card' will contain monthly pooled, agency-level information summarizing clinical data for injured children stratified by race/ethnicity. At month 7 the investigators will also distribute Battalion-level 'Equity Report Cards' to agency leadership and all frontline EMS providers.

SUMMARY:
This trial will assess whether development and sharing of 'Equity Report Cards' focussed on the recognition and treatment of pain for injured children by Emergency Medical Services (EMS) can help decrease disparities by race and ethnicity.

DETAILED DESCRIPTION:
This is a pragmatic trial using an interrupted time-series design. The investigators will collect two years of retrospective data to establish a baseline. At month 2 the investigators will distribute EMS Agency-level 'Equity Report Cards' to both agency leadership and all frontline EMS providers. This 'Equity Report Card' will contain monthly pooled, agency-level information summarizing clinical data for injured children stratified by race/ethnicity. At month 7 the investigators will also distribute Battalion-level 'Equity Report Cards' to agency leadership and all frontline EMS providers. The 'Equity Report Card' will include baseline historical data and a 3-month rolling average for each of the study outcomes. The 'Equity Report Card' will also include an action plan with evidenced based recommendations specifically targeted to improve care.

The outcomes for this study include both process measures (including documentation of pain scores, administration of any analgesia and administration of opiate analgesia) and also patient-centered clinical outcomes (reduction of pain as reported by the patient). These key study outcomes align with performance measures developed by the National EMS Quality Alliance (NEMSQA).

Patient race and ethnicity will be abstracted from the EMS medical record. The investigators will also collect data regarding potential confounding variables including patient age, sex, geographic location of encounter and other dispatch details.

The investigators will conduct an interrupted time series analysis (ITSA) to evaluate the magnitude and statistical significance of the average difference (intercept) and difference between trajectories (slopes) for our 24 month control (T0) and each of the two intervention 5 month time periods (T1 and T2). This will allow the investigators to measure the impact of each additional intervention (EMS agency-level followed by the addition of Battalion-level 'Equity Report Cards').

ELIGIBILITY:
Inclusion Criteria:

* Children less than 18 years old
* Assessed by District of Columbia Fire and Emergency Medical Services (DC FEMS)
* Injury related chief complaint, primary or secondary impression

Exclusion Criteria:

- None

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4000 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in pain | 1 year
  Proportion of children who have a reduction in pain score

SECONDARY OUTCOMES:
Pain score documented | 1 year
  Proportion of children who have a pain score documented by EMS
Any analgesia administered | 1 year
  Proportion of children who have any analgesia administered by EMS
Opiate analgesia administered | 1 year
  Proportion of children who have opiate analgesia administered by EMS

CONTACTS AND LOCATIONS:
Overall Officials: Caleb E Ward, MD, MPH, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No